CLINICAL TRIAL: NCT02756247
Title: Phase Ib Clinical Trial of Buparlisib and Ibrutinib in Mantle Cell Lymphoma, Follicular Lymphoma and Diffuse Large B Cell Lymphoma
Brief Title: A Clinical Trial of Buparlisib and Ibrutinib in Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Janssen Scientific Affairs, LLC (Industry); Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-009
Record Dates: First submitted 2016-04-27; First posted 2016-04-29 (Estimated); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Lymphoma; Mantle Cell Lymphoma; Follicular Lymphoma; Diffuse Large B Cell Lymphoma
Keywords: Buparlisib; BKM120; Ibrutinib; 16-009
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — NVP-BKM120; ibrutinib

ARMS (1):
- Buparlisib and Ibrutinib (Experimental): This is a two stage protocol comprised of a single institution phase Ib dose escalation trial. The first stage is a standard 3+3 phase I dose escalation trial to assess the safety of buparlisib and ibrutinib. The second stage is a single center expansion cohort in MCL, FL and DLBCL respectively evaluating the efficacy of buparlisib and ibrutinib combination.
  Treatment will be with ibrutinib orally daily and buparlisib orally daily. A cycle is defined as 4 weeks of therapy. Therapy will continue until disease progression, intolerable toxicities or death with a maximum duration for 36 cycles, not exceeding 36 months on therapy.
  Interventions: Drug: Buparlisib; Drug: Ibrutinib

INTERVENTIONS:
Drug: Buparlisib
Drug: Ibrutinib

SUMMARY:
The purpose of this study is to find out if the combination of buparlisib and ibrutinib will lead to better treatment results in patients with relapsed or refractory Follicular lymphoma, (FL) Mantle cell lymphoma (MCL) or Diffuse Large B-cell lymphoma (DLBCL). The investigators are using buparlisib and ibrutinib because both drugs seem to block different proteins that allow cancer cells to keep growing. Blocking these proteins may help by making the cancer cells undergo cell death, which will stop uncontrolled tumor growth.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 18 years of age at the time of signing Informed Consent
* Patient is able and willing to adhere to the study visit schedule and other protocol requirements
* Patient has histologically confirmed diagnosis of R/R mantle cell lymphoma, follicular lymphoma or diffuse large B cell lymphoma

  * Diffuse large B cell lymphoma patients has received at least 1 prior regimen and received, declined, or is ineligible for autologous or allogeneic stem cell transplant.
  * Follicular lymphoma patients have received at least 2 lines of therapy.
  * Mantle cell lymphoma patients has received at least 1 line of therapy
  * Allogeneic stem cell transplant recipients be greater than 6 months post transplant, not on immunosuppression for prevention of graft versus host disease for >3 months and without active graft versus host disease are eligible
  * Autologous stem cell transplant recipients must have adequate bone marrow recovery and transfusion independent
  * Transformed histologies are permitted
* Patient has at least one measurable lesion (≥ 2 cm) according to Lugano Classification
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patient has adequate bone marrow and organ function by:

  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L , independent of growth factor support unless with bone marrow involvement for 14 days
  * Platelets ≥100 x 109/L, or ≥50 x 10^9/L if bone marrow involvement and independent of transfusion support for 14 days in either situation
  * Hemoglobin (Hgb) ≥ 9.0 g/dL (no RBC transfusion within past 14 days)
  * Hgb >/= 8.0 g/dL for patients with anemia associated disease
  * International Normalized Ratio (INR) ≤ 1.5
  * Serum Creatinine ≤ 1.5 x upper limit of normal (ULN) or creatinine clearance ≥ 25 mL/min as determined by the Cockcroft-Gault equation or a 24 hour urine collection
  * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ ULN (or ≤3 x ULN if liver involved with disease
  * Total serum bilirubin ≤ ULN (or ≤ 1.5 x ULN if documented hepatic involvement; or total bilirubin ≤ 3 x ULN with direct bilirubin ≤ 1.5 x ULN in patients with documented Gilbert's Syndrome
  * LVEF ≥ 50%
  * Fasting plasma glucose (FPG) ≤ 120mg/dL or ≤ 6.7 mmol/L
  * Hemoglobin A1c ≤ 9%
  * Potassium and calcium (corrected for albumin), within normal limits for the institution, or ≤ Grade 1 if judged not clinically significant by the investigator
* Women of childbearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trial. Men must agree to not donate sperm during and after the study.

  ° For females, these restrictions apply for 1 month after the last dose of study drug. For males, these restrictions apply for 4 months after the last dose of study drug.
* Women of childbearing potential must have a negative serum (beta-human chorionic gonadotropin) or urine pregnancy test at Screening. Women who are pregnant or breastfeeding are ineligible for this study.
* Patient is able to swallow and retain oral medications

Exclusion Criteria:

* Patients previously treated with ibrutinib or PI3K inhibitor
* Patient has a history of non-compliance to medical regimen or inability to grant consent
* Patient has not recovered to Grade 1 or better (except alopecia) from related side effects of any prior antineoplastic therapy.
* Patient is concurrently using other approved or investigational antineoplastic agent
* Patient has had major surgery or a wound that has not fully healed within 4 weeks of starting study drugs.
* Patients who have had chemotherapy or radiotherapy within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 2 weeks earlier
* Patient has evidence of active graft versus host disease (GVHD)
* Patient has active or history of central nervous system (CNS) disease or meningeal involvement.
* Patient has history of stroke or intracranial hemorrhage ≤ 6 months from starting study drugs.
* Patient has a score ≥ 12 on the PHQ-9 questionnaire, selects a response of "1, 2 or 3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9), score ≥ 15 on GAD-7 mood scale.
* Patient has ≥ CTCAE grade 3 anxiety Patient has a medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, homicidal ideation (e.g. risk of doing harm to self or others)
* Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of study drug (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
* Patient has clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification. Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO), unstable angina pectoris, symptomatic pericarditis, QTcF > 480 msec on the screening ECG (using the QTcF formula)
* Patient has a concurrent active malignancy. Malignancies treated with a curative intent with an expected life expectancy ≥ 5 years or a non-competing life expectancy risk are eligible (i.e. adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer, early stage breast cancer, treated prostate cancer or any other cancer from which the patient has been disease free for >/= 3 years).
* Patient with known history of human immunodeficiency virus (HIV), or any uncontrolled active systemic infection.
* Patient has acute viral hepatitis (typically defined by elevated AST/ALT), or a history of chronic or active HBV or HCV infection. HBV infection is defined as having HBsAg and/or HBcAb positive test HBsAg and/or HBcAb positive test detectable HBV DNA levels. HCV infection is defined as detectable HCV RNA levels.
* Patient is currently receiving increasing or chronic treatment (> 5 days) with corticosteroids or another immunosuppressive agent. The following uses of corticosteroids are permitted: single doses; e.g. with standard premedication for taxanes; topical applications (e.g., rash), inhaled sprays (e.g., obstructive airways diseases), eye drops or local injections (e.g., intra-articular); patients requiring chronic therapy with steroids may take no more than 10mg daily of prednisone or equivalent.
* Patient requires treatment with a strong or moderate cytochrome P450 (CYP) 3A4 inhibitors, and inducers, or drugs known to induce Torsades de Pointes and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patients with known bleeding diathesis (e.g. von Willebrand 's disease) or hemophilia
* Patient is currently receiving warfarin or other Vitamin K antagonist. Therapy with heparin, low molecular weight heparin (LMWH), or fondaparinux is allowed. Refer to Section 9.5 for Concomitant medication
* Patients with Child Pugh Class B or C hepatic cirrhosis
* Vaccinated with live attenuated vaccines ≤ 4 weeks from starting study drugs.
* Patients with any life threatening illness, medical condition or organ system dysfunction that in the opinion of the investigator could compromise the subject's safety, interfere with absorption of metabolism of study drugs or put the study outcomes at undue risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2022-10-06 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 1 year
  In the Phase I part the standard 3+3 dose escalation scheme will be used and all disease subtypes will be combined. If none of the initial cohort of 3 has a DLT the dose level will be escalated. If one has a DLT that dose level will be expanded with 3 more patients. Dose escalation will stop if 2 or more DLTs are seen at a dose level. The MTD is defined as the highest dose level at which at most 1 of the 6 patients treated at that level has a DLT. Three dose levels plus a "-1" dose level are planned for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Connie Batlevi, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Stewart CM, Michaud L, Whiting K, Nakajima R, Nichols C, De Frank S, Hamlin PA Jr, Matasar MJ, Gerecitano JF, Drullinsky P, Hamilton A, Straus D, Horwitz SM, Kumar A, Moskowitz CH, Moskowitz A, Zelenetz AD, Rademaker J, Salles G, Seshan V, Schoder H, Younes A, Tsui DWY, Batlevi CL. Phase I/Ib Study of the Efficacy and Safety of Buparlisib and Ibrutinib Therapy in MCL, FL, and DLBCL with Serial Cell-Free DNA Monitoring. Clin Cancer Res. 2022 Jan 1;28(1):45-56. doi: 10.1158/1078-0432.CCR-21-2183. Epub 2021 Oct 6. PMID 34615723
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/